CLINICAL TRIAL: NCT05240898
Title: A Phase 1 Study of RO7623066 Alone and in Combination in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WP45169; KSQ-4279-1101 (Other: KSQ Therapeutics, Inc.)
Record Dates: First submitted 2022-01-26; First posted 2022-02-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — olaparib; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RO7623066 Monotherapy (Dose Escalation) (Experimental): RO7623066 will be administered orally once daily (QD) continuously as monotherapy. Once the maximum tolerated dose (MTD) for RO7623066 monotherapy has been reached this concludes the Dose Escalation phase.
  Interventions: Drug: RO7623066
- RO7623066 + Olaparib (Dose Escalation and Expansion) (Experimental): RO7623066 will be tested in combination with olaparib. Escalating dose levels will be tested until the maximum tolerated dose (MTD), or lower, of RO7623066 is reached or MTD, or lower, of the combination is reached (whichever occurs first). Combination arms can enroll concurrently. Olaparib will be dosed per standard of care (SoC).
  Interventions: Drug: RO7623066; Drug: Olaparib
- RO7623066 + Carboplatin (Dose Escalation and Expansion) (Experimental): RO7623066 will be tested in combination with carboplatin. Escalating dose levels will be tested until the maximum tolerated dose (MTD), or lower, of RO7623066 is reached or MTD, or lower, of the combination is reached (whichever occurs first). Combination arms can enroll concurrently. Carboplatin will be dosed per standard of care (SoC).
  Interventions: Drug: RO7623066; Drug: Carboplatin
- RO7623066 + Olaparib Backfill Cohort (Other): Once safety data has been obtained in the RO7623066 + Olaparib arm during the dose escalation phase, Backfill cohorts will be used to determine the Recommended Dose for Expansion of RO7623066 + Olaparib.
  Interventions: Drug: RO7623066; Drug: Olaparib
- RO7623066 Food Effect Cohort (Other): The effect of food intake on the PK of RO7623066 will be explored at a dose close to the Maximum Tolerated Dose (MTD) and/or at Recommended Phase II Dose (RP2D) or at a relevant dose level for a minimum of 12 participants that have at least one tumor mutation of interest.
  Interventions: Drug: RO7623066

INTERVENTIONS:
Drug: RO7623066 — Administered orally in capsule
  Other Names: KSQ-4279
Drug: Olaparib — Administered orally.
  Dose levels and schedules will be selected based on integration of preclinical data as well as clinical PK, safety, efficacy, and PD/biomarker data (as appropriate) from the dose escalation cohorts.
  Arms: RO7623066 + Olaparib (Dose Escalation and Expansion); RO7623066 + Olaparib Backfill Cohort
Drug: Carboplatin — Administered intravenously.
  Arms: RO7623066 + Carboplatin (Dose Escalation and Expansion)

SUMMARY:
This is a Phase 1 study to assess the safety and clinical activity of RO7623066 alone and in combination in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1 study consisting of 2 parts: Dose Escalation and Expansion to evaluate the safety, tolerability, clinical activity, and pharmacokinetics (PK) Study of RO7623066 as a Monotherapy or in Combination in Patients with Advanced Solid Tumors, and a Food Effect Cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Life expectancy of ≥ 12 weeks
3. Measurable disease or non-measurable disease per RECIST v1.1 in dose escalation and the Food Effect Cohort only; patients in dose expansion and Backfill Cohorts are required to have measurable disease per RECIST v1.1
4. Recovered to ≤ Grade 1 or baseline toxicity (except alopecia) from prior therapy (per NCI-CTCAE v5.0)
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Adequate bone marrow function defined as:

   1. absolute neutrophil count of ≥ 1.5 × 109/L
   2. platelet count of ≥ 100.0 × 109/L
   3. hemoglobin of ≥ 10.0 g/dL (with or without transfusion)
7. Adequate renal function defined as calculated creatinine clearance (Cockcroft- Gault) ≥ 40 mL/min for patients with creatinine levels above institutional normal
8. Adequate hepatic function defined as:

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) unless associated with Gilbert's syndrome
   2. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 × ULN (or ≤ 5 × ULN in patients with liver metastases)
9. Female patients who are women of childbearing potential (WOCP) (defined as physiologically and anatomically capable of becoming pregnant), confirmed of a negative pregnancy test and agreement to the use of a highly effective contraceptive method or at least 2 effective methods at the same time during study treatment period and for up to 3 months after the last dose of study treatment. Male patients must be willing to use effective barrier contraception (ie, condoms) during the study treatment period and for up 3 months after the last dose of study treatment
10. Capable of understanding and complying with protocol requirements
11. Signed and dated institutional review board (IRB)/independent ethics committee (IEC) approved informed consent form (ICF) before any protocol-directed Screening procedures are performed
12. Does not require ongoing treatment with strong or moderate CYP3A4 inhibitors or inducers.
13. Histologically or cytologically confirmed locally advanced (unresectable) or metastatic solid tumors who meet one of the following criteria (dose escalation only):

    1. Relapsed or progressed through standard therapy
    2. Have a disease for which no standard effective therapy exists
    3. Not a candidate for standard effective therapy Note: In men with prostate cancer, baseline testosterone levels must also be ≤ 50 ng/dL (≤ 2.0 nM) and surgical or ongoing medical castration must be maintained throughout the duration of the study

Exclusion Criteria:

1. Prior anticancer treatment including:

   1. Chemotherapy or small molecule-targeted therapy < 2 weeks prior to first dose of study treatment
   2. Any antibody therapy < 5 half-lives from first dose of study treatment (or 4 weeks since last therapy, whichever is the shortest)
   3. Programmed cell death protein-1 or programmed cell death ligand 1 inhibitor therapy < 4 weeks from first dose of study treatment
   4. Invasive surgery requiring general anesthesia < 30 days from first dose of study treatment
   5. Chemotherapy with nitrosoureas or mitomycin C < 45 days from first dose of study treatment
   6. Radiation therapy (including radiofrequency ablation) < 4 weeks prior to initiation of study treatment Note: Prior stereotactic body radiation therapy or local palliative radiation is allowed < 2 weeks prior to first dose of study treatment
2. Ongoing Grade 2 or greater toxicity, except alopecia, related to any prior treatment (ie, chemotherapy, targeted therapy, radiation, or surgery)
3. Prolongation of QT/QTc interval (QTc interval > 480 msec) using the Frederica method of QTc analysis
4. Women who are pregnant or nursing
5. Seropositive for human immunodeficiency virus (HIV) 1 or 2 or acquired immunodeficiency syndrome or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV) (Note: Patients with positive HCV antibody may be eligible if HCV ribonucleic acid [RNA] is undetectable on a quantitative HCV RNA assay, the Medical Monitor is available for advice)
6. Primary malignant brain tumor
7. Symptomatic and/or untreated brain metastases, active leptomeningeal disease, or central nervous system malignant disease requiring steroids or other therapeutic intervention Note: Patients with definitively treated brain metastases will be considered for enrollment after seeking advice from the Medical Monitor and must be clinically stable for ≥ 2 weeks prior to the start of treatment
8. Previous solid organ or hematopoietic cell transplant
9. Need for treatment with steroids at stable doses (> 10 mg prednisone or equivalent per day). Note: Oral steroids up to 10 mg/day, topical, ophthalmic, or inhaled steroid medications are allowed
10. Uncontrolled hypertension > 150/100 mm Hg despite aggressive therapy
11. Concurrent participation in any other investigational therapeutic study
12. History of stroke, transient ischemic attack, unstable angina, or myocardial infarction within 3 months prior to first dose of study treatment
13. Unable to swallow whole tablets or capsules. Nasogastric or gastric-tube (G-tube)administration is not allowed
14. GI disease that would impair ability to swallow, retain, or absorb drug is not allowed
15. Uncontrolled concurrent disease or illness including but not limited to:

    1. Symptomatic congestive heart failure according to New York Heart Association (NYHA) classification, Class III or IV (per NYHA Classification) unstable angina pectoris, or clinically significant cardia arrhythmia
    2. Diabetes mellitus (ie, fasting blood glucose > 220 despite acceptable chronic diabetes therapy)
    3. Psychiatric illness that would limit compliance with study requirements, as determined by the Investigator
16. Other severe, acute, or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or that may interfere with the interpretation of the study results, and in the judgment of the Investigator, would make the patient inappropriate for the study
17. Known hypersensitivity to any component of RO7623066 or excipient
18. History of and/or ongoing adrenal disorder (eg, Cushing's disease, Addison's disease, adrenal gland suppression)
19. Suspected pneumonitis or interstitial lung disease (confirmed radiography or by computed tomography [CT]) or a history of pneumonitis or interstitial lung disease in the last 6 months
20. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, or other cancer for which the patient has been disease-free for at least 2 years
21. Myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML), or baseline features suggestive of MDS or AML on peripheral blood smear or bone marrow biopsy
22. Treatment with strong or moderate CYP3A4 inhibitors or inducers for a period of 5 half-lives of the inhibitor or inducer prior to the first dose of RO7623066.
23. Blood transfusions within 4 weeks prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose (MTD) Measured by the Incidence of Dose Limiting Toxicities (DLTs) | Approximately 4 years 10 months

SECONDARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and change from baseline in laboratory results | Approximately 4 years 10 months
  Assess safety and tolerability
Pharmacokinetics (PK) parameters of RO7623066 | Approximately 4 years 10 months
  PK parameters of RO7623066, including maximum plasma concentration (Cmax), time to Cmax (Tmax), total exposure (area under the concentration-time curve [AUC]), clearance (CL), volume of distribution (Vd), and half-life (T1/2)
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) Investigator assessment | Approximately 4 years 10 months
  Anti-tumor activity
Progression-free survival (PFS) per RECIST v1.1 Investigator assessment | Approximately 4 years 10 months
  Anti-tumor activity
Duration of response (DOR) per RECIST v1.1 Investigator assessment | Approximately 4 years 10 months
  Anti-tumor activity
Time to response (TTR) per RECIST v1.1 Investigator assessment | Approximately 4 years 10 months
  Anti-tumor activity
Overall survival (OS), defined as the date of first dose of study drug to the date of death from any cause | Approximately 4 years 10 months
  Anti-tumor activity
Effect of food on PK parameters | Approximately 4 years 10 months
  PK parameters such as Cmax, Tmax, AUC, and T1/2 for participants who received study treatment who were either in a fed state or in a fasted state.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (15):
  - University of California Irvine Medical Center, Orange, California
  - Yale School of Medicine, New Haven, Connecticut
  - Barbara Ann Karmanos Cancer Institute, Detroit, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics (START) - Midwest Location, Grand Rapids, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic,, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Mary Crowley Medical Research Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No